CLINICAL TRIAL: NCT04668209
Title: Phase II, Randomized, Investigator Initiated Trial to Evaluate Safety and to Explore Clinical Benefit of Silmitasertib (CX-4945) in Patients With Severe Coronavirus Disease 2019 (COVID-19)
Brief Title: Silmitasertib (CX-4945) in Patients With Severe Coronavirus Disease 2019 (COVID-19)
Acronym: CX4945
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After 15 months of active enrollment and a lack of qualifying hospitalized COVID-19 patients, the Sponsor-Investigator, Marilyn Csete Glassberg, MD, decided to terminate recruitment before meeting the stated enrollment objectives.
Sponsor: University of Arizona (Other)
Collaborators: Senhwa Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX4945-AV02-IIT
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-11

CONDITIONS: Coronavirus
Keywords: SARS-CoV-2; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — silmitasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Silmitasertib (Active Comparator): Standard of care / supportive care in combination with Silmitasertib (CX-4945)
  Interventions: Drug: Silmitasertib
- Standard of Care (No Intervention): Standard of care / supportive care

INTERVENTIONS:
Drug: Silmitasertib — Standard of care / best supportive care in combination with CX-4945 1000 mg administered orally, two times a day.
  Other Names: CX-4945
  Arms: Silmitasertib

SUMMARY:
This multi-center, open-label, 2 arm parallel-group, randomized, interventional prospective exploratory study in 40 patients aimed to evaluate safety and explore putative clinical benefits of Silmitasertib 1000 mg BID dose in patients with severe illness caused be SARS-COV-2. This will be a two-arm trial comparing the SOC/best supportive care alone to the SOC/best supportive care with addition of Silmitasertib (allocation ratio 1:1).

DETAILED DESCRIPTION:
This is a phase II multi-center, randomized, open-label, 2 arm parallel-group controlled interventional prospective study of CX-4945 in patients with severe COVID-19. Up to approximately 40 patients will be enrolled into this study. A screening evaluation will occur within 7 days prior to Day 1. All qualified patients will be randomized at Day 1 in a ratio of 1:1 to one of the following two treatment arms:

Arm A: SOC/ best supportive care in combination with CX-4945 1000 mg BID PO or Arm B: SOC/ best supportive care alone The standard of care (SOC) is not pre-specified, may vary among patients, and may include agents with anti-viral activity, such as remdesivir, among others. Investigator discretion is to be applied for any established SOC. Active concomitant treatment with other investigational antivirals or immunomodulators are not permitted Best supportive care is defined as intensive care therapy according to current guidelines, evidence, and best practice, including but not limited to lung protective ventilation, thrombosis prophylaxis, renal replacement therapy when indicated, and access to advanced therapies including extracorporeal membrane oxygenation.

The total duration of the treatment will be 14 days. Patients will be followed up at 28, 45 and 60 days from the start of the treatment. The total duration for each patient in the study (including the screening) will be up to 67 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female adult ≥ 18 years of age
2. Diagnosed/confirmed with COVID-19 by standard RT-PCR assay or equivalent testing within 7 days prior to randomization (Day1).
3. Hospitalized patient with severe illness caused by SARS-CoV-2 (Note: Prior or current use of remdesivir or dexamethasone (SOC) are allowed under the investigator's discretion. Concomitant treatment with other investigational antiviral drugs or immunomodulators are not permitted from Day1 through Day 28)

   Symptoms of severe systemic illness/infection with COVID-19:

   At least 1 of the following: fever, cough, sore throat, malaise, headache, muscle pain, shortness of breath at rest or with exertion, confusion, or symptoms of severe lower respiratory infection including dyspnea at rest or respiratory distress AND Clinical signs indicative of severe systemic illness/infection with COVID-19 At least 1 of the following: RR ≥ 30, HR ≥ 125, SaO2 <93% on room air or requires > 2L oxygen by nasal cannula in order to maintain SaO2 ≥93%
4. Patient (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
5. Adequate hematopoietic capacity, as defined by the following:

   1. Hemoglobin ≥ 9.0 g/dL and not transfusion dependent
   2. Platelets ≥ 100,000/mm3
   3. Absolute neutrophil count ≥ 1500 cells/mm3
6. Adequate hepatic function, as defined by the following:

   1. AST and ALT ≤ 2.5 times upper limit of normal (ULN)
   2. Total bilirubin ≤ 1.5 x ULN
   3. Albumin ≥ 3.0 g/dL
7. Adequate renal function, as defined by the following:

   a. Renal: calculated creatinine clearance >45 mL/min for patients with abnormal, increased creatinine levels (Cockcroft-Gault formula).
8. Ability to take oral medication and be willing to adhere to drug administration and premedication requirements (see Section 6.3) throughout study duration.

Exclusion Criteria:

1. Patient showing signs of respiratory failure necessitating mechanical ventilation
2. Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a man father a child, or a woman become pregnant or suspect she is pregnant while participating in this study, he or she should inform the treating physician immediately.
3. Active or uncontrolled infections other than COVID-19 or with serious illnesses or medical conditions which would not permit the patient to receive study treatment
4. Active or planned concomitant treatment with other investigational antivirals or immunomodulators
5. Chronic diarrhea (excess of 2-3 stools/day above normal frequency)
6. Current use or anticipated need for drugs that are known strong inhibitors or inducers of major CYP enzymes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Banner University Medical Center Tucson, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No
Study results will be published on clinicaltrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from patients hospitalized with diagnosed/confirmed COVID-19 at two academic medical centers between January 2021 and April 2022. The first participant was enrolled on January 21st, 2021, and the last was enrolled in February 2022.
Pre-assignment Details: Of the 31 enrolled participants, 29 met inclusion criteria and were randomized.
Groups:
- Silmitasertib (CX-4945) in Combination With Standard of Care: Standard of care / supportive care in combination with Silmitasertib (CX-4945)
  Participants received Silmitasertib (CX-4945) 1000 mg tablets orally twice a day for 14 days. Participants received supportive care/Standard of Care as assigned by the investigator.
- Standard of Care: Participants received supportive care/Standard of Care.
Period: Overall Study
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Started | 15 | 14
Completed | 8 | 6
Not Completed | 7 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 3 | 4
Not completed — Subject Expired | 2 | 0
Not completed — Withdrawn from study | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (14.72) | 43.9 (13.04) | 46.4 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 15 | 11 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events [Safety and Tolerability]
Description: Adverse Events experienced by the patients from randomization to Day 60 (including vital signs, physical findings, clinical laboratory, and ECG results) as characterized by type, frequency, severity (as graded by Common Terminology Criteria for Adverse Events (CTCAE version 5.0), timing, seriousness, and relationship to study therapy.
Time Frame: Through Day 60
Population: Intent to treat population (all participants assigned to Silmitasertib/Combo, or Standard of Care). The median treatment duration of Silmitasertib was 14 days. The treatment Durations (days) = the last administration date - the first administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 14
Participants
  Experienced Incidence of Treatment Emergent Adverse Events | 10 | 7
  Did not experience Incidence of Treatment Emergent Adverse Events | 5 | 7

2. Secondary Outcome: To Compare Time to Clinical Recovery in CX-4945 Treatment Group Evaluated From Randomization Through Day 28 as Compared to the Control Arm.
Description: Number of days from randomization to discharge, or to alleviation of cough (defined as mild or absent in a patient reported scale of 0=absent, 1=mild, 2=moderate, and 3=severe). Improvement must be sustained for at least 48 hours.
Time Frame: Through Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Silmitasertib | Standard of Care
Number analyzed (Participants) | 15 | 14
Days | 3 (1.5) | 3.4 (1.3)

3. Secondary Outcome: To Compare Time to Clinical Recovery in CX-4945 Treatment Group Evaluated From Randomization Through Day 28 as Compared to the Control Arm.
Description: Number of days from randomization to normalization of fever (defined as <36.6°C from axillary site, or < 37.2°C from oral site or < 37.8°C from rectal or tympanic site), normalization of respiratory rate (< 24 bpm while breathing room air), resolution of hypoxia (defined as SpO2 ≥ 93% in room air or P/F ≥ 300 mmHg). All these improvements must be sustained for at least 48 hours.
Time Frame: Through hospital discharge, an average of 28 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 14
Days | 6 (4.1) | 5.1 (2.9)

4. Secondary Outcome: To Compare Time to Clinical Recovery in CX-4945 Treatment Group Evaluated From Randomization Through Day 28 as Compared to the Control Arm.
Description: Number of days from randomization to the first day on which the subject satisfies one of the following three categories from the ordinal NIAID 8- point Clinical Progression Outcomes scale collected daily from randomization through Day 28:
  Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; Not hospitalized, limitation on activities and/or requiring home oxygen; Not hospitalized, no limitations on activities.
Time Frame: Through Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 14
Days | 7.3 (4.6) | 6 (3.3)

5. Secondary Outcome: To Compare Changes in Clinical Status of Patients Enrolled to CX-4945 Treatment Arm as Compared to the Control Arm at Day 14 and Day 28.
Description: Difference in percentage of subjects with clinical recovery compared at Day 14 and Day 28.
Time Frame: Assessed on Day 14 and Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 14
Participants
  Day 14 | 13 | 13
  Day 28 | 13 | 13

6. Secondary Outcome: To Compare Changes in Clinical Status of Patients Enrolled to CX-4945 Treatment Arm as Compared to the Control Arm at Day 14 and Day 28.
Description: Percentage of Participants at Each Clinical Status at Day 14 and Day 28 assessed by using the ordinal NIAID 8- point Clinical Progression Outcomes scale (Scale ranges from 1 (Death) to 8 (Not hospitalized, no limitations on activities)
Time Frame: Through Day 28
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 11 | 9
Participants
  Day 14: Death | 0 | 0
  Day 14: Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | 1 | 2
  Day 14: Hospitalized, on non-invasive ventilation or high flow oxygen devices | 1 | 1
  Day 14: Hospitalized, requiring supplemental oxygen | 2 | 0
  Day 14: Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 0 | 0
  Day 14: Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 0 | 0
  Day 14: Not hospitalized, limitation on activities and/or requiring home oxygen | 5 | 2
  Day 14: Not hospitalized, no limitations on activities | 2 | 4
  Day 28: number analyzed (Participants) | 10 | 6
  Day 28: Death | 2 | 0
  Day 28: Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | 0 | 2
  Day 28: Hospitalized, on non-invasive ventilation or high flow oxygen devices | 0 | 0
  Day 28: Hospitalized, requiring supplemental oxygen | 0 | 0
  Day 28: Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 0 | 0
  Day 28: Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 0 | 0
  Day 28: Not hospitalized, limitation on activities and/or requiring home oxygen | 4 | 1
  Day 28: Not hospitalized, no limitations on activities | 4 | 3

7. Secondary Outcome: To Evaluate Preliminary Evidence of Anti-viral Activity of CX-4945 as Compared to the Control Arm.
Description: Difference in proportions of patients with conversion of positive RT-PCR to negative RT-PCR as assessed at Day 1, Day 8, Day 14 and Day 28.
Time Frame: Assessed at Day 1, Day 8, Day 14 and Day 28
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 12
Participants
  Day 1: Positive | 15 | 12
  Day 1: Negative | 0 | 0
  Day 8: number analyzed (Participants) | 11 | 6
  Day 8: Positive | 8 | 4
  Day 8: Negative | 3 | 2
  Day 14: number analyzed (Participants) | 9 | 5
  Day 14: Positive | 4 | 3
  Day 14: Negative | 5 | 2
  Day 28: number analyzed (Participants) | 5 | 5
  Day 28: Positive | 1 | 0
  Day 28: Negative | 4 | 5

8. Secondary Outcome: To Evaluate Preliminary Evidence of Anti-viral Activity of CX-4945 as Compared to the Control Arm.
Description: Changes in chest imaging from Screening to Day 5 or 14
Time Frame: Through Day 14
Population: No data collected for this outcome analysis.
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Days Hospitalized
Description: Days of hospitalization from randomization through Day 28
Time Frame: Through Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 12 | 10
Days | 10.1 (8.4) | 11.7 (19.7)

10. Secondary Outcome: To Evaluate Changes in IL-6 Level
Description: IL-6 level
Time Frame: Assessed on Days 1, 4, 8, 11, and 14
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 13 | 11
Participants
  Day 1: Abnormal: High | 5 | 6
  Day 1: Abnormal: Low | 0 | 0
  Day 1: Normal | 8 | 5
  Day 1: Unable to determine | 0 | 0
  Day 4: number analyzed (Participants) | 9 | 11
  Day 4: Abnormal: High | 4 | 4
  Day 4: Abnormal: Low | 0 | 0
  Day 4: Normal | 4 | 7
  Day 4: Unable to determine | 1 | 0
  Day 8: number analyzed (Participants) | 8 | 5
  Day 8: Abnormal: High | 5 | 3
  Day 8: Abnormal: Low | 0 | 0
  Day 8: Normal | 1 | 2
  Day 8: Unable to determine | 2 | 0
  Day 11: number analyzed (Participants) | 8 | 6
  Day 11: Abnormal: High | 7 | 5
  Day 11: Abnormal: Low | 0 | 0
  Day 11: Normal | 1 | 1
  Day 11: Unable to determine | 0 | 0
  Day 14: number analyzed (Participants) | 9 | 5
  Day 14: Abnormal: High | 6 | 5
  Day 14: Abnormal: Low | 0 | 0
  Day 14: Normal | 3 | 0
  Day 14: Unable to determine | 0 | 0

11. Secondary Outcome: To Evaluate Changes in CRP
Description: CRP level
Time Frame: Assessed on Days 1, 4, 8, 11, and 14
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 13
Participants
  Day 1: Abnormal: High | 12 | 13
  Day 1: Abnormal: Low | 0 | 0
  Day 1: Normal | 3 | 0
  Day 1: Unable to determine | 0 | 0
  Day 4: number analyzed (Participants) | 12 | 12
  Day 4: Abnormal: High | 8 | 8
  Day 4: Abnormal: Low | 0 | 0
  Day 4: Normal | 4 | 4
  Day 4: Unable to determine | 0 | 0
  Day 8: number analyzed (Participants) | 10 | 6
  Day 8: Abnormal: High | 8 | 3
  Day 8: Abnormal: Low | 0 | 0
  Day 8: Normal | 2 | 3
  Day 8: Unable to determine | 0 | 0
  Day 11: number analyzed (Participants) | 10 | 5
  Day 11: Abnormal: High | 8 | 5
  Day 11: Abnormal: Low | 0 | 0
  Day 11: Normal | 1 | 0
  Day 11: Unable to determine | 1 | 0
  Day 14: number analyzed (Participants) | 9 | 5
  Day 14: Abnormal: High | 6 | 4
  Day 14: Abnormal: Low | 0 | 0
  Day 14: Normal | 2 | 1
  Day 14: Unable to determine | 1 | 0

12. Secondary Outcome: To Evaluate Changes in LDH
Description: LDH level
Time Frame: Assessed on Days 1, 4, 8, 11, and 14
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 14 | 13
Participants
  Day1: Abnormal: High | 13 | 13
  Day1: Abnormal: Low | 1 | 0
  Day1: Normal | 0 | 0
  Day1: Unable to determine | 0 | 0
  Day 4: number analyzed (Participants) | 12 | 12
  Day 4: Abnormal: High | 12 | 11
  Day 4: Abnormal: Low | 0 | 0
  Day 4: Normal | 0 | 1
  Day 4: Unable to determine | 0 | 0
  Day 8: number analyzed (Participants) | 11 | 5
  Day 8: Abnormal: High | 11 | 4
  Day 8: Abnormal: Low | 0 | 1
  Day 8: Normal | 0 | 0
  Day 8: Unable to determine | 0 | 0
  Day 11: number analyzed (Participants) | 10 | 6
  Day 11: Abnormal: High | 9 | 6
  Day 11: Abnormal: Low | 0 | 0
  Day 11: Normal | 1 | 0
  Day 11: Unable to determine | 0 | 0
  Day 14: number analyzed (Participants) | 9 | 5
  Day 14: Abnormal: High | 8 | 2
  Day 14: Abnormal: Low | 0 | 0
  Day 14: Normal | 1 | 2
  Day 14: Unable to determine | 0 | 1

13. Secondary Outcome: To Evaluate Changes in CPK
Description: CPK level
Time Frame: Assessed on Days 1, 4, 8, 11, and 14
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 13 | 13
Participants
  Day 1: Abnormal: High | 1 | 1
  Day 1: Abnormal: Low | 4 | 2
  Day 1: Normal | 8 | 10
  Day 1: Unable to determine | 0 | 0
  Day 4: number analyzed (Participants) | 12 | 12
  Day 4: Abnormal: High | 2 | 0
  Day 4: Abnormal: Low | 4 | 4
  Day 4: Normal | 6 | 8
  Day 4: Unable to determine | 0 | 0
  Day 8: number analyzed (Participants) | 11 | 6
  Day 8: Abnormal: High | 1 | 0
  Day 8: Abnormal: Low | 6 | 1
  Day 8: Normal | 3 | 5
  Day 8: Unable to determine | 1 | 0
  Day 11: number analyzed (Participants) | 10 | 7
  Day 11: Abnormal: High | 1 | 0
  Day 11: Abnormal: Low | 2 | 3
  Day 11: Normal | 7 | 4
  Day 11: Unable to determine | 0 | 0
  Day 14: number analyzed (Participants) | 10 | 5
  Day 14: Abnormal: High | 1 | 0
  Day 14: Abnormal: Low | 1 | 2
  Day 14: Normal | 8 | 3
  Day 14: Unable to determine | 0 | 0

14. Secondary Outcome: To Evaluate Changes in Ferritin
Description: Ferritin level
Time Frame: Assessed on Days 1, 4, 8, 11, and 14
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 14 | 13
Participants
  Day 1: Abnormal: High | 13 | 8
  Day 1: Abnormal: Low | 0 | 0
  Day 1: Normal | 1 | 5
  Day 1: Unable to determine | 0 | 0
  Day 4: number analyzed (Participants) | 12 | 11
  Day 4: Abnormal: High | 11 | 7
  Day 4: Abnormal: Low | 0 | 0
  Day 4: Normal | 1 | 3
  Day 4: Unable to determine | 0 | 1
  Day 8: number analyzed (Participants) | 11 | 5
  Day 8: Abnormal: High | 9 | 4
  Day 8: Abnormal: Low | 0 | 0
  Day 8: Normal | 1 | 1
  Day 8: Unable to determine | 1 | 0
  Day 11: number analyzed (Participants) | 10 | 7
  Day 11: Abnormal: High | 8 | 5
  Day 11: Abnormal: Low | 0 | 0
  Day 11: Normal | 2 | 2
  Day 11: Unable to determine | 0 | 0
  Day 14: number analyzed (Participants) | 10 | 5
  Day 14: Abnormal: High | 6 | 3
  Day 14: Abnormal: Low | 1 | 0
  Day 14: Normal | 3 | 1
  Day 14: Unable to determine | 0 | 1

15. Secondary Outcome: To Evaluate Changes in D-dimer
Description: D-dimer level
Time Frame: Assessed on Days 1, 4, 8, 11, and 14
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 14 | 13
Participants
  Day 1: Abnormal: High | 10 | 8
  Day 1: Abnormal: Low | 0 | 0
  Day 1: Normal | 2 | 3
  Day 1: Unable to determine | 2 | 2
  Day 4: number analyzed (Participants) | 12 | 12
  Day 4: Abnormal: High | 10 | 10
  Day 4: Abnormal: Low | 0 | 0
  Day 4: Normal | 2 | 2
  Day 4: Unable to determine | 0 | 0
  Day 8: number analyzed (Participants) | 11 | 6
  Day 8: Abnormal: High | 9 | 5
  Day 8: Abnormal: Low | 0 | 0
  Day 8: Normal | 1 | 1
  Day 8: Unable to determine | 1 | 0
  Day 11: number analyzed (Participants) | 10 | 6
  Day 11: Abnormal: High | 9 | 5
  Day 11: Abnormal: Low | 0 | 0
  Day 11: Normal | 1 | 1
  Day 11: Unable to determine | 0 | 0
  Day 14: number analyzed (Participants) | 10 | 5
  Day 14: Abnormal: High | 8 | 4
  Day 14: Abnormal: Low | 0 | 0
  Day 14: Normal | 0 | 1
  Day 14: Unable to determine | 2 | 0

16. Secondary Outcome: Number of Days of Supplemental Oxygen Use
Description: Days of supplemental oxygen (if applicable) from randomization through day 28
Time Frame: Through Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 14
Days | 4.8 (4.6) | 4.2 (3.2)

17. Secondary Outcome: All-cause Mortality Status
Description: The number of deaths occurred in each treatment group from randomization through Day 60
Time Frame: Through Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 14
Participants
  Death - Yes | 2 | 2
  Death - No | 13 | 12

18. Secondary Outcome: Number of Days of On-invasive Ventilation/High Flow Oxygen
Description: Days of non-invasive ventilation/high flow oxygen (if applicable) from randomization through day 28
Time Frame: Through Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 14
Days | 2.1 (4.1) | 1.9 (2.9)

19. Secondary Outcome: Number of Days of Invasive Mechanical Ventilation/ECMO
Description: Days of invasive mechanical ventilation/ECMO (if applicable) from randomization through Day 28.
Time Frame: Through Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 14
Days | 1.9 (5.3) | 3 (7.7)

20. Secondary Outcome: Number of Patients Returned to Room Air
Description: Number of patients returned to room air after randomization through Day 14 or Day 28.
Time Frame: Through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 15 | 14
Participants
  Day 14: Return to room air: Yes | 12 | 10
  Day 14: Return to room air: No | 3 | 4
  Day 28: Return to room air: Yes | 12 | 10
  Day 28: Return to room air: No | 3 | 4

21. Secondary Outcome: Change in Pulse Oxygen Saturation
Description: Change in pulse oxygen saturation (SpO2) from randomization to Day 4, 8, 11, 14 and 28
Time Frame: Days 4, 8, 11, 14, and 28
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin saturation
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 13 | 12
percentage of hemoglobin saturation
  Day 4 | 0.5 (3.4) | -1.1 (1.8)
  Day 8: number analyzed (Participants) | 12 | 7
  Day 8 | 1.3 (3.3) | 0.3 (3.6)
  Day 11: number analyzed (Participants) | 10 | 8
  Day 11 | -0.4 (4.8) | -0.5 (5.6)
  Day 14: number analyzed (Participants) | 10 | 9
  Day 14 | -0.5 (3.9) | -1.8 (8.8)
  Day 28: number analyzed (Participants) | 7 | 6
  Day 28 | 1.7 (2.6) | 1.7 (3.7)

22. Secondary Outcome: Number of Thrombosis Events
Description: Number of documented venous thromboembolism (VTE), arterial thrombosis (stroke, myocardial infarction, other) and microthrombosis events from randomization through Day 28
Time Frame: Through Day 28
Population: No data collected for this outcome analysis.
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Changes in EQ-D5-5L
Description: The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). Higher values indicate worse outcomes, while lower indicate better outcomes. The subscales are combined to compute a total score and averaged to produce the mean and SD.
  Changes in EQ-D5-5L (used as an indicator of symptom improvement) from randomization to Day 8, 14 and 28
Time Frame: Days randomization, 8, 14 and 28
Population: Missing data explains the discrepancy in the total analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 9
score on a scale
  Day 8 Mobility score | -1 (1.6) | -1.7 (1.2)
  Day 14 Mobility score: number analyzed (Participants) | 9 | 7
  Day 14 Mobility score | -1.1 (1.6) | -1.7 (1.5)
  Day 28 Mobility score: number analyzed (Participants) | 9 | 5
  Day 28 Mobility score | -1.4 (1.9) | -2.6 (1.1)
  Day 8 Self-care score | -1.2 (1.6) | -2.1 (2.6)
  Day 14 Self-care score: number analyzed (Participants) | 9 | 7
  Day 14 Self-care score | -1.1 (1.8) | -3 (1.7)
  Day 28 Self-care score: number analyzed (Participants) | 9 | 5
  Day 28 Self-care score | -1.3 (1.7) | -2.8 (1.3)
  Day 8 Usual activities score | -2.3 (1.6) | -0.7 (2.2)
  Day 14 Usual activities score: number analyzed (Participants) | 9 | 7
  Day 14 Usual activities score | -2.3 (1.6) | -1.4 (1.4)
  Day 28 Usual activities score: number analyzed (Participants) | 9 | 5
  Day 28 Usual activities score | -2.6 (1.6) | -1.4 (1.3)
  Day 8 Pain/discomfort score | 0.3 (1.1) | -0.8 (1)
  Day 14 Pain/discomfort score: number analyzed (Participants) | 9 | 7
  Day 14 Pain/discomfort score | -0.2 (0.4) | -0.3 (1.3)
  Day 28 Pain/discomfort score: number analyzed (Participants) | 9 | 5
  Day 28 Pain/discomfort score | -0.3 (0.7) | -0.2 (1.3)
  Day 8 Anxiety/depression score | 0 (0.8) | 0.1 (0.6)
  Day 14 Anxiety/depression score: number analyzed (Participants) | 9 | 7
  Day 14 Anxiety/depression score | -0.2 (0.7) | -0.1 (1.2)
  Day 28 Anxiety/depression score: number analyzed (Participants) | 9 | 5
  Day 28 Anxiety/depression score | 0 (0.5) | -0.2 (1.1)

ADVERSE EVENTS:
Time Frame: Day 60.
Description: Adverse Events experienced by patients from randomization to Day 60 (including vital signs, physical findings, clinical laboratory, and ECG results) as characterized by type, frequency, severity (as graded by Common Terminology Criteria for Adverse Events (CTCAE version 5.0), timing, seriousness, and relationship to study therapy.
Arm/Group | Silmitasertib (CX-4945) in Combination With Standard of Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/15 | 2/14
Serious Adverse Events (participants affected / at risk) | 3/15 | 2/14
Other Adverse Events (participants affected / at risk) | 10/15 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silmitasertib (CX-4945) in Combination With Standard of Care (N=15) | Standard of Care (N=14)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnea worsened (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Premature atrial contractions (Cardiac disorders) | 1 | 1
Acute hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silmitasertib (CX-4945) in Combination With Standard of Care (N=15) | Standard of Care (N=14)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Premature atrial contractions (Cardiac disorders) | 0 | 1
Bloody diarrhea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 2
Diarrhea worsened (Gastrointestinal disorders) | 1 | 0
Loose stools (Gastrointestinal disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
Weakness (General disorders) | 0 | 1
Pilonidal cyst worsened (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 1
Decrease appetite (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Leg Pain Bilateral (Musculoskeletal and connective tissue disorders) | 1 | 0
Anosmia (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression worsened (Psychiatric disorders) | 0 | 1
Acute hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnea worsened (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Worsening hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis anal (Skin and subcutaneous tissue disorders) | 1 | 0
Sweating (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
After 15 months of active enrollment and a lack of qualifying hospitalized COVID-19 patients, the Sponsor-Investigator, Marilyn Csete Glassberg, MD, decided to terminate recruitment before meeting the stated enrollment objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT04668209/Prot_SAP_002.pdf
  • Informed Consent Form (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT04668209/ICF_003.pdf